CLINICAL TRIAL: NCT04733885
Title: Evaluation of the Effects of Electrical Stimulation in Women With Pelvic Organ
Brief Title: Electrical Stimulation in Women With Pelvic Organ Prolapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Collaborators: Ankara Yildirim Beyazıt University (Other); Necmettin Erbakan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KaratayZK
Record Dates: First submitted 2021-01-24; First posted 2021-02-02 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2021-01

CONDITIONS: Pelvic Organ Prolapse
Keywords: pelvic organ prolapse; electrical stimulation
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Electric Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electrical Stimulation group (Experimental): ES and lifestyle advice have been applied ES application will be done 3 days a week for 8 weeks, 20 minutes. An informative brochure with lifestyle advice will be provided for both groups.
  Interventions: Device: Experimental
- Sham Electric Stimulation group (Sham Comparator): Sham ES and lifestyle advice have been applied Sham ES application will be done 3 days a week for 8 weeks, 20 minutes. An informative brochure with lifestyle advice will be provided for both groups.
  Interventions: Device: Control

INTERVENTIONS:
Device: Experimental — Current application will be made in the frequency range of 20-50 Hz. The Chattanooga (Intelect Neo) device with interfering current will be used for treatment, vacuum electrodes will be made in the form of 4 pole application. Two electrodes to the outside of the inguinal ligament, the other two electrodes will be placed on the upper inner part of the thigh.ES applications will be performed in the supine position with head and knee pillow supported.
  Other Names: Electrical Stimulation
  Arms: Electrical Stimulation group
Device: Control — The Chattanooga (Intelect Neo) device with interfering current will be used for treatment, vacuum electrodes will be made in the form of 4 pole application. Two electrodes to the outside of the inguinal ligament, the other two electrodes will be placed on the upper inner part of the thigh. The same device used in ES application to the sham group will be attached to the patients, however, active ES will not be issued from the device and only vacuum will turn on. ES applications will be performed in the supine position with head and knee pillow supported.
  Other Names: Sham Electrical Stimulation
  Arms: Sham Electric Stimulation group

SUMMARY:
The aim of this study is to search the effects of electrical stimulation on clinical symptoms such as pelvic floor muscle strength, stage of POP, symptoms of pelvic floor, quality of life and sexual function in women with pelvic organ prolapse (POP)

DETAILED DESCRIPTION:
This study is planned as a prospective, sham radomized controlled study. Individuals who volunteered to participate in the study, complying with the inclusion criteria and signed the consent paper will be randomly allocated into ES and Sham ES groups.

The study includes women aged 18-65 diagnosed with staged 1-2 POP by the physician.All patients were evaluated by the same doctor who performed the POP-Q measurement, who was blinded to the baseline results. The treatment of patients will be given by the same therapist. Measurements will be made 3 times at baseline (before treatment), interim period (4th week) and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Being in the age range of 18-65 ,
* Having stage1-2 symptomatic prolapse according to the POP-Q system,
* Being a volunteer and literate

Exclusion Criteria:

* Being pregnant,
* being stage 3-4 prolapse, Those whose evaluation parameters are missing and who do not regularly participate,
* Inadequate understanding and cooperation in treatment and evaluation parameters,
* Have malignant disease, urinary infection,
* accompanying neurological disease, diabetes mellitus and cardiopathy with complications,
* have electronic and metal implant, loss of sensation, sacral peripheral nerve lesion
* Patients with at least one of the kidney failure requiring hemodialysis

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 26 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
The prolapse stage will be measured with Simplified POP-Q | Change from baseline prolapse stage at 4 weeks and 8 weeks
  The measurements are taken when the Valsalva maneuver is performed while the patient is in the dorsal lithotomy position. According to the reference point of the hymen, It is measured at a total of 4 points: cervix, posterior fornix, anterior and posterior vaginal wall. The stage of prolapse is graded.
  Stage 0: There is no prolapse. Stage 1: The most distal part of the prolapse is more than 1 cm above the prolapse.
  Stage 2: The most distal part of the prolapse, between 1 cm above and 1 cm below the prolapse Stage 3: The most distal part of the prolapse protrudes more than 1 cm below the prolapse.
  Stage 4: Complete eversion of the lower genital tract

SECONDARY OUTCOMES:
Pelvic floor muscle strength will be measured measured with PFX Perineometer device(Cardio Design Pty Ltd, Australia) | Change from baseline Pelvic floor muscle strength at 4 weeks and 8 weeks
  Indicators of this measuring device range from 0-12 kilo Pascal (kPa). During the measurement, The patient whose perineometer sensor is placed in her vagina, will be asked to relax and then to tighten the sensor strongly. The difference between the first and last value in the perineometer is the contraction strength. This evaluation will be repeated three times and averaged and recorded.
The pelvic organ prolapse symptoms will be assessed by Pelvic Organ Prolapse Symptom Score(POP-SS). | Change from baseline the pelvic organ prolapse symptoms at 4 weeks and 8 weeks
  Pelvic Organ Prolapse Symptom Score (POP-SS) consists of 7 questions whose answers are scored between 0 and 5. The total score ranges from 0 to 28. The higher the score, the higher the severity of POP symptoms.
The pelvic organ prolapse symptoms severity will be assessed by the Pelvic Floor Distress Inventory (PFDI-20) . | Change from baseline the pelvic organ prolapse symptoms severity at 4 weeks and 8 weeks
  The PFDI comprises three subscales: the Pelvic Organ Prolapse Distress Inventory-6, the ColoRectal-Anal Distress Inventory-8 and the Urinary Distress Inventory-6. The scores range from 0 to l00 for the all subscales. Higher scores signifying severe symptom.
Patients' quality of life will be assessed using the Prolapse Quality of Life Scale (P-QOL). | Change from baseline quality of life at 4 weeks and 8 weeks
  The scale consists of 9 fields and 20 questions. The first question is general health perception, the second question is the effect of urogenital prolapse on the quality of life, the 3rd and 4th questions are role limitations, the 5th and 6th questions are physical limitations, the 7th and 8th questions are social limitations, 9-11. questions on interpersonal relationships, 12-14. questions ask emotions, questions 15 and 16 examine sleep / energy influence, and questions 16 and 20 examine severity. The score ranges from 0-100, with a higher score indicating poor quality of life.
Patients' sexual function will be assessed by the Pelvic Organ Prolapse/Incontinence Sexual Function Questionnaire-12 (PISQ-12) | Change from baseline sexual function at 4 weeks and 8 weeks
  This survey, consisting of 12 questions, includes 3 subtitles.This survey, consisting of 12 questions, includes 3 subtitles. 1-4. Questions are emotional, 5-9. questions are physical, 10-12. questions constitute subheadings containing partner dependent areas (range 0-48, with higher scores indicating better sexual functioning).

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No